CLINICAL TRIAL: NCT04526535
Title: Prognostic Value of Lung Ultrasound in ST Segment Elevation Acute Myocardial Infarction (LUS-AMI)
Acronym: LUS-AMI
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Institut Hospital del Mar d'Investigacions Médiques (Unknown); Hospital Vall d'Hebron (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ECO-2019-105
Record Dates: First submitted 2020-07-24; First posted 2020-08-26 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Acute Myocardial Infarction; Heart Failure
Keywords: Lung Ultrasound
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No B-lines: Patients with no significant B lines in the lung ultrasound at first 24 hours after acute myocardial infarction (any field with 3 or more B-lines)
  Interventions: Diagnostic Test: Lung ultrasound
- B lines: Patients with significant B lines in the lung ultrasound at first 24 hours after acute myocardial infarction (3 or more B-lines in at least one lung field)
  Interventions: Diagnostic Test: Lung ultrasound

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — Lung ultrasound performed with a portable device with an 8 zones protocol within the first 24 hours after and ST-segment elevation acute myocardial infarction

SUMMARY:
The purpose of this study is to asses the prognostic value of lung ultrasound in patients with ST-segment elevation acute myocardial infarction.

DETAILED DESCRIPTION:
LUS-AMI is an observational cohort prospective study that evaluates the prognostic value of lung ultrasound, specifically the number of B-lines, performed within the first 24 hours after and ST-segment elevation acute myocardial infarction, by an independent operator blinded to clinical outcomes and off-line analysis by another independent operator also blinded to clinical outcomes.

The primary outcome during hospitalization was a composite of clinically significant acute HF, cardiogenic shock, or death from any cause after LUS was performed. New-onset atrial fibrillation, acute renal injury (Acute Kidney Injury Network ≥ 1), and need for ventilatory support (invasive or non-invasive) during hospitalization were also analyzed as secondary outcomes.

The primary outcome during follow-up is one year after STEMI is a composite of any cause mortality, hospitalization secondary to cardiovascular disease (aborted sudden cardiac arrest, acute coronary syndrome, heart failure or stroke) or need for urgent coronary revascularization.

Secondary outcomes are new onset heart failure during hospitalization, acute kidney injury during hospitalization, new-onset atrial fibrillation/flutter during hospitalization, need of ventilatory support during hospitalization and new-onset clinically relevant arrhythmia (atrial fibrillation, atrial flutter, ventricular tachycardia, ventricular fibrillation) during follow-up. A short-term follow-uo (30 days after prior PCI) will be also performed to analyze a combined endpoint of death from any cause or hospitalization due to acute HF or new acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adults (more than 18 years) admitted with confirmed ST-segment elevation acute myocardial infarction (STEMI).

Exclusion Criteria:

* Absence of coronary artery disease and myocardial injury (false positive)
* Non interpretable lung ultrasound
* Severe lung disease (fibrosis, severe COPD, pleural disease, lobectomy or pneumonectomy)
* Acute respiratory distress syndrome
* Pneumonia or SDRA at admission or during hospitalization
* Follow-up inability
* Hemodialysis therapy previous to admission
* Life expectancy less than 6 months secondary to extracardiac pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults admitted with STEMI during 1 year in three terciary centers who meet inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Primary combined outcome: incidence of any cause mortality or hospitalization secondary to cardiovascular cause. | Up to 12 months since revascularization and LUS performance.
  Combined outcome of: mortality from any cause, readmission due to cardiovascular cause (aborted sudden cardiac arrest, acute coronary syndrome, heart failure or stroke) or the need for urgent coronary revascularization at a 12-month follow-up since prior revascularization.

SECONDARY OUTCOMES:
Combined endpoint during hospitalization: death or acute heart failure (congestive HF or cardiogenic shock) in STEMI Killip I patients. | During hospitalization due to prior STEMI, after revascularization and LUS performance.
  Acute congestive heart failure, defined as the presence of three conditions: 1) dyspnea at rest; 2) peripheral oxygen saturation (SpO2) <90% or need for oxygen to maintain adequate SpO2; and 3) presence of crackles or elevated natriuretic peptides (NTproBNP >450 pg/ml <50 years-old, >900 50-75y, >1800 >75 years-old). Cardiogenic shock was defined according to current guidelines as systolic blood pressure <90 mm Hg for at least 30 minutes or the need for supportive measures to maintain systolic blood pressure ≥90 mm Hg) despite adequate filling status with clinical and laboratory evidence of end-organ hypoperfusion. This outcome will be analyzed only in patients without signs of HF at admission (Killip I).
Combined endpoint in a short follow-up: heart failure, acute coronary syndrome or death, | Up to 30 days since prior revascularization
  Composite of readmission for acute HF or new ACS (hospitalization or >24 hours of stay in the Emergency Department) or death from any cause.
Acute renal injury during hospitalization | During hospitalization due to prior STEMI, after revascularization and LUS performance.
  Acute Kidney Injury Network (AKIN) criteria I, II or III or hemodialysis requirement
Development of atrial fibrilation/flutter during hospitalization | During hospitalization due to prior STEMI, after revascularization and LUS performance.
  New-onset atrial fibrillation or atrial flutter during hospitalization in patients without prior history of these arrhythmias.
Ventilatory support during hospitalization | During hospitalization due to prior STEMI, after revascularization and LUS performance.
  Need of ventilatory support (invasive or non-invasive mechanical ventilation) during hospitalization.
Development of arrhythmias during follow-up | Up to 12 months
  New-onset atrial fibrillation, atrial flutter, sustained ventricular tachycardia or ventricular fibrillation during hospitalization and during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carreras-Mora, MD., Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (2):
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Farré N, Fort A, Tizón-Marcos H, et al. Epidemiology of heart failure in myocardial infarction treated with primary angioplasty: Analysis of the Codi IAM registry. REC: CardioClinics 2019;54:41-49.
- [Result] Araujo GND, Marques F, Scolari F, et al. Comparison of Lung Ultrasound and Killip Classification in Patients with St-Segment Elevation Myocardial Infarction Submitted to Coronary Angiography. J Am Coll Cardiol 2019;73:182.
- [Result] Lichtenstein DA. BLUE-protocol and FALLS-protocol: two applications of lung ultrasound in the critically ill. Chest. 2015 Jun;147(6):1659-1670. doi: 10.1378/chest.14-1313. PMID 26033127
- [Result] Pivetta E, Goffi A, Lupia E, Tizzani M, Porrino G, Ferreri E, Volpicelli G, Balzaretti P, Banderali A, Iacobucci A, Locatelli S, Casoli G, Stone MB, Maule MM, Baldi I, Merletti F, Cibinel GA, Baron P, Battista S, Buonafede G, Busso V, Conterno A, Del Rizzo P, Ferrera P, Pecetto PF, Moiraghi C, Morello F, Steri F, Ciccone G, Calasso C, Caserta MA, Civita M, Condo' C, D'Alessandro V, Del Colle S, Ferrero S, Griot G, Laurita E, Lazzero A, Lo Curto F, Michelazzo M, Nicosia V, Palmari N, Ricchiardi A, Rolfo A, Rostagno R, Bar F, Boero E, Frascisco M, Micossi I, Mussa A, Stefanone V, Agricola R, Cordero G, Corradi F, Runzo C, Soragna A, Sciullo D, Vercillo D, Allione A, Artana N, Corsini F, Dutto L, Lauria G, Morgillo T, Tartaglino B, Bergandi D, Cassetta I, Masera C, Garrone M, Ghiselli G, Ausiello L, Barutta L, Bernardi E, Bono A, Forno D, Lamorte A, Lison D, Lorenzati B, Maggio E, Masi I, Maggiorotto M, Novelli G, Panero F, Perotto M, Ravazzoli M, Saglio E, Soardo F, Tizzani A, Tizzani P, Tullio M, Ulla M, Romagnoli E; SIMEU Group for Lung Ultrasound in the Emergency Department in Piedmont. Lung Ultrasound-Implemented Diagnosis of Acute Decompensated Heart Failure in the ED: A SIMEU Multicenter Study. Chest. 2015 Jul;148(1):202-210. doi: 10.1378/chest.14-2608. PMID 25654562
- [Result] Lichtenstein D, Goldstein I, Mourgeon E, Cluzel P, Grenier P, Rouby JJ. Comparative diagnostic performances of auscultation, chest radiography, and lung ultrasonography in acute respiratory distress syndrome. Anesthesiology. 2004 Jan;100(1):9-15. doi: 10.1097/00000542-200401000-00006. PMID 14695718
- [Result] Coiro S, Rossignol P, Ambrosio G, Carluccio E, Alunni G, Murrone A, Tritto I, Zannad F, Girerd N. Prognostic value of residual pulmonary congestion at discharge assessed by lung ultrasound imaging in heart failure. Eur J Heart Fail. 2015 Nov;17(11):1172-81. doi: 10.1002/ejhf.344. Epub 2015 Sep 29. PMID 26417699
- [Result] Platz E, Lewis EF, Uno H, Peck J, Pivetta E, Merz AA, Hempel D, Wilson C, Frasure SE, Jhund PS, Cheng S, Solomon SD. Detection and prognostic value of pulmonary congestion by lung ultrasound in ambulatory heart failure patients. Eur Heart J. 2016 Apr 14;37(15):1244-51. doi: 10.1093/eurheartj/ehv745. Epub 2016 Jan 26. PMID 26819225
- [Result] Rivas-Lasarte M, Alvarez-Garcia J, Fernandez-Martinez J, Maestro A, Lopez-Lopez L, Sole-Gonzalez E, Pirla MJ, Mesado N, Mirabet S, Fluvia P, Brossa V, Sionis A, Roig E, Cinca J. Lung ultrasound-guided treatment in ambulatory patients with heart failure: a randomized controlled clinical trial (LUS-HF study). Eur J Heart Fail. 2019 Dec;21(12):1605-1613. doi: 10.1002/ejhf.1604. Epub 2019 Oct 31. PMID 31667987
- [Result] Januzzi JL, van Kimmenade R, Lainchbury J, Bayes-Genis A, Ordonez-Llanos J, Santalo-Bel M, Pinto YM, Richards M. NT-proBNP testing for diagnosis and short-term prognosis in acute destabilized heart failure: an international pooled analysis of 1256 patients: the International Collaborative of NT-proBNP Study. Eur Heart J. 2006 Feb;27(3):330-7. doi: 10.1093/eurheartj/ehi631. Epub 2005 Nov 17. PMID 16293638
- [Result] Platz E, Jhund PS, Girerd N, Pivetta E, McMurray JJV, Peacock WF, Masip J, Martin-Sanchez FJ, Miro O, Price S, Cullen L, Maisel AS, Vrints C, Cowie MR, DiSomma S, Bueno H, Mebazaa A, Gualandro DM, Tavares M, Metra M, Coats AJS, Ruschitzka F, Seferovic PM, Mueller C; Study Group on Acute Heart Failure of the Acute Cardiovascular Care Association and the Heart Failure Association of the European Society of Cardiology. Expert consensus document: Reporting checklist for quantification of pulmonary congestion by lung ultrasound in heart failure. Eur J Heart Fail. 2019 Jul;21(7):844-851. doi: 10.1002/ejhf.1499. Epub 2019 Jun 19. PMID 31218825
- [Result] Ye XJ, Li N, Li JH, Wu WJ, Li AL, Li XL. B-lines by lung ultrasound predict heart failure in hospitalized patients with acute anterior wall STEMI. Echocardiography. 2019 Jul;36(7):1253-1262. doi: 10.1111/echo.14420. Epub 2019 Jul 9. PMID 31287587
- [Result] Araujo GN, Silveira AD, Scolari FL, Custodio JL, Marques FP, Beltrame R, Menegazzo W, Machado GP, Fuchs FC, Goncalves SC, Wainstein RV, Leiria TL, Wainstein MV. Admission Bedside Lung Ultrasound Reclassifies Mortality Prediction in Patients With ST-Segment-Elevation Myocardial Infarction. Circ Cardiovasc Imaging. 2020 Jun;13(6):e010269. doi: 10.1161/CIRCIMAGING.119.010269. Epub 2020 Jun 15. PMID 32536197
- [Derived] Carreras-Mora J, Vidal-Burdeus M, Rodriguez-Gonzalez C, Simon-Ramon C, Rodriguez-Sotelo L, Sionis A, Giralt-Borrell T, Martinez-Membrive MJ, Izquierdo-Marquisa A, Farre N, Cainzos-Achirica M, Tizon-Marcos H, Garcia-Picart J, Mila-Pascual L, Vaquerizo-Montilla B, Rivas-Lasarte M, Ribas-Barquet N. Lung Ultrasound in the Acute Phase of ST-Segment-Elevation Acute Myocardial Infarction: 1-Year Prognosis and Improvement in Risk Prediction. J Am Heart Assoc. 2024 Nov 5;13(21):e035688. doi: 10.1161/JAHA.124.035688. Epub 2024 Oct 29. PMID 39470045